CLINICAL TRIAL: NCT05101720
Title: Ultrasound Guided Axillary Access vs Standard Fluoroscopic Technique for Cardiac Lead Implantation
Brief Title: Ultrasound Guided Axillary Access vs Standard Fluoroscopic Technique for Cardiac Lead Implantation: ZEROFLUOROAXI TRIAL
Acronym: ZEROFLUOROAXI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Bertini, MD, PhD, Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE-AVEC 555/2021/Sper/AOUFe
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Arrhythmias, Cardiac; Venous Puncture; Implantable Defibrillator User; Pacemaker Complication; Vascular Access Complication; Fluoroscopy; Adverse Effect
Keywords: pacemaker; ICD; arrhythmias; Cardiac Implantable Electronic Device; Vascular access; Venous puncture; Ultrasound; Fluoroscopy
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Axillary Access (Experimental): Direct visualization of axillary vein with ultrasound will be obtained and used as a guidance for venous puncture.
  Interventions: Procedure: Ultrasound Guided Axillary Venous Access
- Fluoroscopic Guided Axillary Access (Active Comparator): Standard technique: using the intersection of the lateral borders of the second and third rib as a radiological landmarks.
  Interventions: Procedure: Fluoroscopy-Guided Axillary Venous Access

INTERVENTIONS:
Procedure: Ultrasound Guided Axillary Venous Access — Direct visualization of axillary vein will be obtained with ultrasound sterile linear probe.
  Arms: Ultrasound Guided Axillary Access
Procedure: Fluoroscopy-Guided Axillary Venous Access — Fluoroscopic landmarks will be used and axillary venous puncture will be performed without ultrasound
  Arms: Fluoroscopic Guided Axillary Access

SUMMARY:
Single center, randomized trial (1:1 fashion) to asses the safety and the feasibility of the ultrasound guided venous puncture vs standard fluoroscopic technique in patients undergoing pacemaker or implantable cardioverter-defibrillator implantations.

DETAILED DESCRIPTION:
Rationale: axillary, cephalic and subclavian venous accesses are commonly used in pacemaker and implantable cardioverter defibrillator implantations. Axillary puncture and cephalic vein surgical cutdown are both recommended in international guidelines due to low risk of pneumothorax and chronic lead complications. Sometimes cephalic vein is not available. Today axillary puncture is performed under fluoroscopic view and some complications still exist with this venous access as pneumothorax and arterial puncture. Axillary vein direct visualization can be obtained with standard venography or with ultrasound. With direct visualization and puncture of the axillary vein under ultrasound guidance venography with radiocontrast could be avoided. Less radiation exposure for patient and operator and direct visualization of the needle are possible with lower periprocedural complications using ultrasound. Despite the great interest for ultrasound guided axillary puncture up today we have few data on its feasibility. Our hypothesis is that ultrasound guided axillary access is more safe and more feasible than the standard fluoroscopic technique.

We decided to enroll all the patients undergoing standard transvenous pacemaker or cardioverter implantable defibrillator. We randomize the patients with 1:1 fashion to axillary venous access under fluoroscopic guidance or to ultrasound guided axillary venous access.

Obiectives: to asses safety, feasibility of the ultrasound guided venous puncture.

Main Endpoint: composite of pneumothorax, pocket hematoma, arterial puncture, pocket or device infection, hemothorax at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Need of a standard transvenous pacemaker or implantable cardioverter defibrillator implantations
* Age > 18 years

Exclusion Criteria:

* Leadless pacemaker or subcutaneous ICD

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Composite of pneumothorax, pocket hematoma, arterial puncture, pocket or device infection, hemothorax at 30 days. | One month after index procedure
  Composite of pneumothorax, pocket hematoma, arterial puncture, pocket or device infection, hemothorax at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertini, MD, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Vitali F, Malagu M, Bianchi N, De Raffele M, Manfrini M, Gibiino F, Boccadoro A, Azzolini G, Balla C, Bertini M. Ultrasound-Guided Venous Axillary Access Versus Standard Fluoroscopic Technique for Cardiac Lead Implantation: ZEROFLUOROAXI Randomized Trial. JACC Clin Electrophysiol. 2024 Mar;10(3):554-565. doi: 10.1016/j.jacep.2023.11.020. Epub 2024 Jan 17. PMID 38243998